CLINICAL TRIAL: NCT02294448
Title: Population Pharmacokinetic Modeling of Qishe Pill in Three Major TCM-defined Constitutional Types of Healthy Chinese Subjects: Study Protocol for a Phase I Clinical Trial
Brief Title: PopPK Profile of Qishe Pill: Study Protocol for a Phase I Clinical Trial
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Cui xuejun, Vice director, Shanghai University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PopPK profile of Qishe Pill
Record Dates: First submitted 2014-09-11; First posted 2014-11-19 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Individuality; Narrative Medicine
Keywords: Cervical radiculopathy; Neck pain; Qishe pill; raditional Chinese medicine; healthy Chinese subject; Population Pharmacokinetics; Personalized Medicine; Individualized Medicine
MeSH Terms: conditions — Narrative Medicine; Radiculopathy; Neck Pain | interventions — qishe

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- cohort 1 (Experimental): Qishe Pill（Shanghai Sundise Traditional Chinese Medicine Co., Ltd, China） in low dosage(3.75mg)
  Interventions: Drug: Qishe Pill
- cohort 2 (Experimental): Qishe Pill（Shanghai Sundise Traditional Chinese Medicine Co., Ltd, China) in medial dosage(7.5mg)
  Interventions: Drug: Qishe Pill
- cohort 3 (Experimental): Qishe Pill（Shanghai Sundise Traditional Chinese Medicine Co., Ltd, China）in high dosage(15mg)
  Interventions: Drug: Qishe Pill

INTERVENTIONS:
Drug: Qishe Pill — Qishe Pill is a thin 0.15 g film-coated pill, composed of processed Radix Astragali, Muscone, Szechuan Lovage Rhizome, Radix Stephaniae Tetrandrae, Ovientvine, and Calculus Bovis Artifactus, which should be taken orally with water (240mL) after a minimum 10-hour fast

SUMMARY:
Qishe Pill (Shanghai Sundise Traditional Chinese Medicine Co., Ltd, China), composed of processed Radix Astragali, Muscone, Szechuan Lovage Rhizome, Radix Stephaniae Tetrandrae, Ovientvine, and Calculus Bovis Artifactus, has been developed and spread in use into clinical settings in 2009. As individualization has become the trend of modern medicine, a personalized medicine of Qishe Pill should be documented and practiced with various patients according to the ancient TCM system, a classification of personalized constitution type, which has been established to determine predisposition and prognosis to diseases as well as therapy and life-style administration. Therefore, we describe the population pharmacokinetic profile of Qishe Pill and compare its extent of metabolism in the 3 major Constitution Type (Qi-Deficiency, Yin-Deficiency and Blood-Stasis) to address major challenges of individualized and standardized Traditional Chinese Medicine into clinical practice.

DETAILED DESCRIPTION:
With the greatly increased morbidity of neck pain, it brought a large challenge to some optimal therapies for various situations in population at a given time based on their demographic, physiological and pathological characteristics. Chinese proprietary herbal medicines, as a kind of Complementary and Alternative Medicine (CAM), are usually developed from some well-established and long-standing recipes and formulated as tablets or capsules for commerce, convenience or palatability. Although these advantage mentioned, a good quantification and a strict standardization in detail are still need to be improved for individualized implementation in therapeutic strategies. Based on the YQHY decoction (Yi-Qi Hua-Yu Decoction, tonify Qi and promoting circulation and removing stasis), Qishe Pill (Shanghai Sundise Traditional Chinese Medicine Co., Ltd, China) has been developed and spread in use into clinical settings in 2009. As individualization has become the trend of modern medicine, a personalized medicine of Qishe Pill should be documented and practiced with various patients according to the ancient TCM system, a classification of personalized constitution type, which has been established to determine predisposition and prognosis to diseases as well as therapy and life-style administration. Therefore, we describe the population pharmacokinetic profile of Qishe Pill and compare its extent of metabolism in the 3 major Constitution Type (Qi-Deficiency, Yin-Deficiency and Blood-Stasis) to address major challenges of individualized and standardized Traditional Chinese Medicine into clinical practice.

ELIGIBILITY:
Inclusion

* Aged 20-35
* 18.5 kg/m2 ≤Body mass index (BMI) <23 kg/m2
* TCM-constitutionally typed as either the 3 major type

Exclusion

* History of impaired fasting glucose or diabetes mellitus (past history of diabetes or fasting blood glucose at screening ≥100 mg/dl)
* History of liver disease (hepatitis, hepatic cirrhosis) or hepatic dysfunction (AST or ALT at screening ≥40 U/L)
* History of renal dysfunction (creatinine at screening ≥1.2 mg/dl)
* History of heart disease (heart failure, angina pectoris, myocardial infarction, arrhythmia)
* History of malignant tumor
* Having digestive disorders that can interfere with normal absorption of standard diet (gastritis, gastric ulcer, duodenitis, duodenal ulcer, etc.)
* Smoking during the recent 3 months
* Alcohol consumption 3 or more times a week during the recent 3 months
* Women who were pregnant, intended to become pregnant, or breast- feeding
* Medicated during the recent month for therapeutic or prophylactic purposes
* Participating in another clinical trial

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-12 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Plasma concentration of Qishe Pill | Dosing(0 hour)
  5 ml blood samples for pharmacokinetic analysis
Plasma concentration of Qishe Pill | 15 min after dosing
  5 ml blood samples for pharmacokinetic analysis
Plasma concentration of Qishe Pill | 30 min after dosing
  5 ml blood samples for pharmacokinetic analysis
Plasma concentration of Qishe Pill | 45 min after dosing
  5 ml blood samples for pharmacokinetic analysis
Plasma concentration of Qishe Pill | 60 min after dosing
  5 ml blood samples for pharmacokinetic analysis
Plasma concentration of Qishe Pill | 90 min after dosing
  5 ml blood samples for pharmacokinetic analysis
Plasma concentration of Qishe Pill | 120 min after dosing
  5 ml blood samples for pharmacokinetic analysis
Plasma concentration of Qishe Pill | 150 min after dosing
  5 ml blood samples for pharmacokinetic analysis
Plasma concentration of Qishe Pill | 180 min after dosing
  5 ml blood samples for pharmacokinetic analysis
Plasma concentration of Qishe Pill | 240 min after dosing
  5 ml blood samples for pharmacokinetic analysis
Plasma concentration of Qishe Pill | 360 min after dosing
  5 ml blood samples for pharmacokinetic analysis
Plasma concentration of Qishe Pill | 480 min after dosing
  5 ml blood samples for pharmacokinetic analysis
Plasma concentration of Qishe Pill | 600 min after dosing
  5 ml blood samples for pharmacokinetic analysis
Plasma concentration of Qishe Pill | 720 min after dosing
  5 ml blood samples for pharmacokinetic analysis
Plasma concentrations of Qishe Pill | 1440 min after dosing
  5 ml blood samples for pharmacokinetic analysis
Plasma concentration of Qishe Pill | 2160 min after dosing
  5 ml blood samples for pharmacokinetic analysis
Plasma sampling of Qishe Pill for pharmacokinetic analysis | 2880 min after dosing
  5 ml blood samples for pharmacokinetic analysis
Vital signs | Dosing(0 hour)
  body temperature, heart rate and blood pressure
Vital signs | 180 min after dosing
  body temperature, heart rate and blood pressure
Vital signs | 720 min after dosing
  body temperature, heart rate and blood pressure
Vital signs | 1440 min after dosing
  body temperature, heart rate and blood pressure
Vital signs | 2160 min after dosing
  body temperature, heart rate and blood pressure
Vital signs | 2880 min after dosing
  body temperature, heart rate and blood pressure
ECG monitoring | Dosing(0 hour)
  Electrocardiograms (ECGs)
ECG monitoring | 180 min after dosing
  Electrocardiograms (ECGs)
ECG monitoring | 720 min after dosing
  Electrocardiograms (ECGs)
ECG monitoring | 1440 min after dosing
  Electrocardiograms (ECGs)
ECG monitoring | 2160 min after dosing
  Electrocardiograms (ECGs)
ECG monitoring | 2880 min after dosing
  Electrocardiograms (ECGs)
Number of Participants with Adverse Events | Day 1 of drug administration and blood sampling
  The investigators will assess all clinical AEs according to the Medical Dictionary for Regular Activities criteria, in terms of intensity (mild, moderate, or severe), duration, outcome and relationship to the study drug.
Number of Participants with Adverse Events | Day 2 of drug administration and blood sampling
  The investigators will assess all clinical AEs according to the Medical Dictionary for Regular Activities criteria, in terms of intensity (mild, moderate, or severe), duration, outcome and relationship to the study drug.
Number of Participants with Adverse Events | Day 3 of drug administration and blood sampling
  The investigators will assess all clinical AEs according to the Medical Dictionary for Regular Activities criteria, in terms of intensity (mild, moderate, or severe), duration, outcome and relationship to the study drug.
Number of Participants with Adverse Events | 4 days after drug administration and blood sampling
  Subjects will be requested to return to the study unit 4 d after drug administration and blood sampling for a follow-up visit.
Peak Plasma Concentration (Cmax) of Qishe Pill in low dosage | 4 days after drug administration and blood sampling
  The maximum plasma concentration
Peak Plasma Concentration (Cmax) of Qishe Pill in medial dosage | 4 days after drug administration and blood sampling
  The maximum plasma concentration
Peak Plasma Concentration (Cmax) of Qishe Pill in high dosage | 4 days after drug administration and blood sampling
  The maximum plasma concentration
The Time to Peak Plasma Concentration (Tmax) of Qishe Pill in low dosage | 4 days after drug administration and blood sampling
  The time to maximum concentration
The Time to Peak Plasma Concentration (Tmax) of Qishe Pill in medial dosage | 4 days after drug administration and blood sampling
  The time to maximum concentration
The Time to Peak Plasma Concentration (Tmax) of Qishe Pill in high dosage | 4 days after drug administration and blood sampling
  The time to maximum concentration
Area under the Plasma Concentration versus Time Curve (AUC) of Qishe Pill in low dosage | 4 days after drug administration and blood sampling
  The area under the plasma concentration-time curve (AUC) will be calculated using the linear trapezoidal rule.
Area under the Plasma Concentration versus Time Curve (AUC) of Qishe Pill in medial dosage | 4 days after drug administration and blood sampling
  The area under the plasma concentration-time curve (AUC) will be calculated using the linear trapezoidal rule.
Area under the Plasma Concentration versus Time Curve (AUC) of Qishe Pill in high dosage | 4 days after drug administration and blood sampling
  The area under the plasma concentration-time curve (AUC) will be calculated using the linear trapezoidal rule.
The distribution volume (DF) of Qishe Pill in low dosage | 4 days after drug administration and blood sampling
  The distribution volume (DF) will be calculated by Dose/AUC/ke. ke is the elimination rate constant.
The distribution volume (DF) of Qishe Pill in medial dosage | 4 days after drug administration and blood sampling
  The distribution volume (DF) will be calculated by Dose/AUC/ke. ke is the elimination rate constant.
The distribution volume (DF) of Qishe Pill in high dosage | 4 days after drug administration and blood sampling
  The distribution volume (DF) will be calculated by Dose/AUC/ke. ke is the elimination rate constant.

SECONDARY OUTCOMES:
Deep phenotyping with genomics and functional genomics approaches | Dosing(0 hour)
  3 ml blood samples for genomic variants analysis. The cytochrome P450 gene family, such as CYP1A1, CYP1A2, CYP2D6, CYP2C9, CYP2C19, CYP2E1, CYP3A4 and CYP3A5 , etc, will be chosen as the target objective.
Deep phenotyping with genomics and functional genomics approaches | 2880 min after dosing
  3 ml blood samples for genomic variants analysis. The cytochrome P450 gene family, such as CYP1A1, CYP1A2, CYP2D6, CYP2C9, CYP2C19, CYP2E1, CYP3A4 and CYP3A5 , etc, will be chosen as the target objective.

OTHER OUTCOMES:
The Constitution in Chinese Medicine Questionnaire (CCMQ) | During screening in the recuitment
  Two qualified traditional Chinese medical doctors licensed by the Chinese government determine the constitution according to CCMQ
The Constitution in Chinese Medicine Questionnaire (CCMQ) | 2880 min after dosing
  Two qualified traditional Chinese medical doctors licensed by the Chinese government determine the constitution according to CCMQ
Laboratory measures and clinical assessment | During screening in the recuitment
  These parameters including blood count, electrolytes, renal and liver function parameters, blood lipids, age, gender, history of smoking, blood pressure, weight (kg), and height (meters) will be obtained for all subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Yong-jun Wang, Dr., Principal Investigator — Longhua Hospital
Locations (1):
- Longhua Hospital, Shanghai University of TCM, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Aker PD, Gross AR, Goldsmith CH, Peloso P. Conservative management of mechanical neck pain: systematic overview and meta-analysis. BMJ. 1996 Nov 23;313(7068):1291-6. PMID 8942688
- [Background] Cui X, Trinh K, Wang YJ. Chinese herbal medicine for chronic neck pain due to cervical degenerative disc disease. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD006556. doi: 10.1002/14651858.CD006556.pub2. PMID 20091597
- [Background] Wang Q. Classification of the nine basic TCM constitutional type and based expression and diagnosis. Journal of Beijing University of Traditional Chinese medicine. 2005.1-8
- [Background] Liu Mei, Zhang N, Wang YJ, Shi Q. Purification process research of major compound in Qishe Pill as Astragalus. Acta Chinese Medicine and Pharmacology. 2006(34):14-16.
- [Background] Zhang YQ, Liu XH, Zhang N, Liu M. Quality standard research of Qishe Pill. Lishizhen Med Mater Med Res. 2008(19): 977-979.
- [Background] Liu M, Zhang N, Wang YJ, Zhang YQ, Zhou CJ. Technology research of Qishe Pill, a new medicine for cervical spondylosis. Lishizhen Med Mater Med Res. 2010(21):176-179.
- [Background] Ge JR, Wang HM, Meng CX, Tong PJ. Effects of Qishe Pill, a compound traditional Chinese herbal medicine, on cervical radiculopathy: a randomized controlled trial for Phase III. Chinese Journal of New Drugs and Clinical. 2014(7):56-58.
- [Background] Johnson CL, Fulwood R, Abraham S, Bryner JD. Basic data on anthropometric measurements and angular measurements of the hip and knee joints for selected age groups 1-74 years of age. Vital Health Stat 11. 1981 Apr;(219):1-68. No abstract available. PMID 15806754
- [Background] Makela M, Heliovaara M, Sievers K, Impivaara O, Knekt P, Aromaa A. Prevalence, determinants, and consequences of chronic neck pain in Finland. Am J Epidemiol. 1991 Dec 1;134(11):1356-67. doi: 10.1093/oxfordjournals.aje.a116038. PMID 1755449
- [Background] Bovim G, Schrader H, Sand T. Neck pain in the general population. Spine (Phila Pa 1976). 1994 Jun 15;19(12):1307-9. doi: 10.1097/00007632-199406000-00001. PMID 8066508
- [Background] van der Donk J, Schouten JS, Passchier J, van Romunde LK, Valkenburg HA. The associations of neck pain with radiological abnormalities of the cervical spine and personality traits in a general population. J Rheumatol. 1991 Dec;18(12):1884-9. PMID 1795327
- [Background] Hsu H-Y: 1986 Oriental MateriaMedica. Long Beach, CA: Oriental Healing Arts Institute; 1986.
- [Background] Zhu YB, Wang Q, Xue HS, Origasa H. Preliminary assessment on performance of constitution in Chinese medicine questionnaire. ZhongGuo Lin Chuang Kang Fu 2006; 10 (3): 15-17.
- [Background] FDA/CDER. Guidance for industry estimating the maximum safe starting dose in initial clinical trials for therapeutics in adult healthy volunteers; 2005, http://www.fda.gov/downloads/drugs/guidance-complianceregulatoryinformation/guidances/ucm078932.pdf.
- [Background] van Gerven J, Bonelli M. Commentary on the EMA Guideline on strategies to identify and mitigate risks for first-in-human and early clinical trials with investigational medicinal products. Br J Clin Pharmacol. 2018 Jul;84(7):1401-1409. doi: 10.1111/bcp.13550. Epub 2018 May 30. No abstract available. PMID 29451320
- [Background] Choo V. WHO reassesses appropriate body-mass index for Asian populations. Lancet. 2002 Jul 20;360(9328):235. doi: 10.1016/S0140-6736(02)09512-0. No abstract available. PMID 12133671
- [Background] Sheiner LB, Beal SL. Evaluation of methods for estimating population pharmacokinetics parameters. I. Michaelis-Menten model: routine clinical pharmacokinetic data. J Pharmacokinet Biopharm. 1980 Dec;8(6):553-71. doi: 10.1007/BF01060053. PMID 7229908
- [Background] Sheiner LB, Beal SL. Evaluation of methods for estimating population pharmacokinetic parameters. II. Biexponential model and experimental pharmacokinetic data. J Pharmacokinet Biopharm. 1981 Oct;9(5):635-51. doi: 10.1007/BF01061030. PMID 7334463
- [Background] Sheiner LB, Beal SL. Evaluation of methods for estimating population pharmacokinetic parameters. III. Monoexponential model: routine clinical pharmacokinetic data. J Pharmacokinet Biopharm. 1983 Jun;11(3):303-19. doi: 10.1007/BF01061870. PMID 6644555
- [Background] Feng Y, Pollock BG, Coley K, Marder S, Miller D, Kirshner M, Aravagiri M, Schneider L, Bies RR. Population pharmacokinetic analysis for risperidone using highly sparse sampling measurements from the CATIE study. Br J Clin Pharmacol. 2008 Nov;66(5):629-39. doi: 10.1111/j.1365-2125.2008.03276.x. Epub 2008 Jul 31. PMID 18771484
- [Background] Zhang WJ, Hufnagl P, Binder BR, Wojta J. Antiinflammatory activity of astragaloside IV is mediated by inhibition of NF-kappaB activation and adhesion molecule expression. Thromb Haemost. 2003 Nov;90(5):904-14. doi: 10.1160/TH03-03-0136. PMID 14597987
- [Derived] Sun YL, Hou T, Liu SF, Zhang ZL, Zhang N, Yao M, Yang L, Shi Q, Cui XJ, Wang YJ. Population pharmacokinetic modeling of the Qishe pill in three major traditional Chinese medicine-defined constitutional types of healthy Chinese subjects: study protocol for a randomized controlled trial. Trials. 2015 Feb 26;16:64. doi: 10.1186/s13063-015-0568-6. PMID 25885543